CLINICAL TRIAL: NCT03900338
Title: Intestinal Microbiota and Its Relationship With Vascular Structure and Function and Cardiovascular Risk, Phase I (MIVAS Study)
Brief Title: Intestinal Microbiota and Arterial Stiffness
Acronym: MIVAS
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: GRS 1820/B/18
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Arterial Stiffness; Dysbiosis
Keywords: pulse wave velocity; intestinal microbiota; cardiovascular disease; short chain fatty acids; multicentric study
MeSH Terms: conditions — Dysbiosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PWV>10: Patients with PWV > 10 (SSphygmoCor) in two different measurements
- PWV<10: Patients with PWV < 10 (SphygmoCor) in two different measurements

SUMMARY:
This is an observational case-control study which objective is to analyse differences in intestinal microbiota between patients with and without arterial stiffness, measured by pulse wave velocity. It will take place in two different research units located in Portugal and Spain.

DETAILED DESCRIPTION:
Aim: analyse differences in intestinal microbiota between patients with and without arterial stiffness, measured by pulse wave velocity.

Design and setting: An observational case-control study. Study population: The investigators will select 324 subjects, between 30 to 75 years-old, from a database that combine data from four different studies: Triple A, Early vascular Aging (EVA) and Improving interMediAte Risk management (MARK) that took place in the Research Unit of La Alamedilla Primary Care Center, and Guimarães/ Vizela Study promoted by the Life and Health Sciences Research Institute in Minho University.

Measurements: 162 Cases will be defined by a Carotid-femoral Pulse Wave Velocity (cf-PWV)>10 mm/s determined using the SphygmoCor System. 162 controls will be selected by the propensity score. The composition of the gut microbiome in faecal samples will be determined by ribosomal ribonucleic acid (16S rRNA) gene sequencing. Other measurements: demographic data, lifestyle assessment (physical activity, adherence to the Mediterranean diet, alcohol and tobacco consumption). Anthropometric Variables: Weight, body composition by bioimpedance, size, body mass index (BMI), waist and hip perimeter, peripheral and central arterial pressure. Analysis of structure and vascular function and organ lesions target: pulse wave velocity, cardio-ankle vascular index and ankle-brachial index; Intimal median carotid thickness, central and peripheral rate of increase, renal and cardiac organic lesion. Blood analysis: short chain fatty acids, total bile acids, ursodeoxycholic acid

ELIGIBILITY:
Inclusion Criteria:

• Patients with more than 40 years old who agree to participate in the study and do not meet any of the exclusion criteria.

Exclusion Criteria:

* Participants who are in terminal condition,
* Participants with a history of cardiovascular disease (ischaemic heart disease or stroke, peripheral arterial disease or Heart Failure),
* People with diabetes,
* diagnosed renal failure in terminal stages (glomerular filtration rate below 30%),
* chronic inflammatory disease or acute inflammatory process in the past 3 months.
* Patients treated with oestrogens, testosterone or growth hormone,

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will select 324 subjects, between 40 to 75 years-old, from a database that combine data from four different studies: Triple A, EVA and Mark that took place in the Research Unit of La Alamedilla Primary Care Center, and Guimarães/ Vizela Study promoted by the Life and Health Sciences Research Institute in Minho University.
  The 162 cases with a pathologic pulse wave velocity will be randomly selected, each of this subjects will be matched to an individual with the same or similar propensity score. Each one of these subjects will go through a PWV study to confirm that they're in the right group.
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | 1 year
  Measurement by SphygmoCor System (meters/seg)

SECONDARY OUTCOMES:
Cardio ankle vascular index | 1 year
  Measurement by Vasera device 2000 (not units)
Carotid intima-media thickness | 1 year
  Measurement by Ultrasonography (Sonosite Micromax) (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia-Ortiz, Study Director — rimary Care Research Unit - The Alamedilla Center for Health; Rita Salvado Martins, Principal Investigator — rimary Care Research Unit - The Alamedilla Center for Health; Pedro Guimaraes Cunha, Study Director — Life and Health Sciences Research Institute in Minho University
Locations (2):
- Life and Health Sciences Research Institute in Minho University, Braga, Portugal
- Primary Care Research Unit - The Alamedilla Center for Health, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salvado R, Lugones-Sanchez C, Santos-Minguez S, Gonzalez-Sanchez S, Quesada JA, Benito R, Rodriguez-Sanchez E, Gomez-Marcos MA, Guimaraes-Cunha P, Hernandez-Rivas JM, Mira A, Garcia-Ortiz L, Mivas Investigators. Sex Differences in Gut Microbiota and Their Relation to Arterial Stiffness (MIVAS Study). Nutrients. 2024 Dec 27;17(1):53. doi: 10.3390/nu17010053. PMID 39796488
- [Derived] Salvado R, Santos-Minguez S, Agudo-Conde C, Lugones-Sanchez C, Cabo-Laso A, M feminine Hernandez-Sanchez J, Benito R, Rodriguez-Sanchez E, Gomez-Marcos MA, Hernandez-Rivas JM, Guimaraes Cunha P, Garcia-Ortiz L, Investigators M. Gut microbiota composition and arterial stiffness measured by pulse wave velocity: case-control study protocol (MIVAS study). BMJ Open. 2021 Feb 11;11(2):e038933. doi: 10.1136/bmjopen-2020-038933. PMID 33574140